CLINICAL TRIAL: NCT02750527
Title: Pediatric Population Screening for Type 1 Diabetes and Familial Hypercholesterolemia in Lower Saxony, Germany
Acronym: Fr1dolin
Status: Completed | Type: Observational
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Responsible Party: Principal Investigator, Olga Kordonouri, Prof. Dr., Kinderkrankenhaus auf der Bult
Other Study IDs: H-Fr1dolin-01
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Type 1 Diabetes; Familial Hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a Pilot/ feasibility study for a population-based Screening in all children 2 to 6 years in Lower Saxony, Germany during the compulsory (U7 (from the age of 2) U7a, U8, U9) routine check-ups and any voluntary visits to the pediatricians office.

DETAILED DESCRIPTION:
The Fr1dolin-Study will be presented to the parents of ca. 320,000 children living in Lower Saxony, Germany. The recruitment of subjects, collection of written consent, the capillary blood sample and the screening questionnaire will be done by the registered pediatricians in their local medical practices.

After study enrolment 200 µl of capillary blood are be taken from the subject and are sent pseudo-anonymized to the lab. LDL-C and the diabetes-associated antibodies are identified. Based on the results a second blood sample will be required. In case of pre-type-1 diabetes or signs for a familial hypercholesterolemia the pediatrician will be informed. He will contact the parents and discuss the further procedure in cooperation with the study center.

In case of a positive result by measuring diabetes-related antibodies and LDL-C the goal of this trial is to advise and educate the families appropriate and to treat them if necessary. In addition families should have the possibility to participate in prevention trials.

All data will be registered in a study database.

Follow-up pre-type 1 diabetes:

During the first year, follow-up will be performed after 6 and 12 months and thereafter annually until the age of 12 years or up to 6 months after the clinical onset of type 1 diabetes.

Follow-up familial hypercholesterolemia:

During the first year, follow-up will be performed after 6 and 12 months and thereafter annually until the age of 12 years.

ELIGIBILITY:
Inclusion Criteria:

* Children living in Lower Saxony (primary residence)
* Age between 2 and 6 years (both included)
* Written consent by at least one parent / legal representative
* Willingness to deliver 200 µl of capillary blood
* Willingness to complete a questionnaire
* Willingness to participate to the follow-up visits

Exclusion Criteria:

• none

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: According to the Federal Statistical Office (31.12.2014) 320.000 children in the age of 2 to 6 years are living in lower Saxony, Germany. Based on the Fr1da experience a participation rate of 25-35 % is expected. The current estimated prevalence of FH und T1D of 1:300 leads to the expected number of 450 newly identified cases of FH and T1D in each case in the period of 18 months. Additional subjects with FH would be identified by cascade screening.
Sampling Method: Probability Sample
Enrollment: 13049 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
number of familial hypercholesterolemia or pre-type-1-diabetes | 18 month
  identification of patients/ families with familial hypercholesterolemia or pre-type-1 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Olga Kordonouri, MD, Principal Investigator — Kinder- und Jugendkrankenhaus AUF DER BULT

IPD SHARING:
Plan to Share IPD: No